CLINICAL TRIAL: NCT04366648
Title: Study on the Safety, Tolerability and Pharmacokinetics of Single and Multiple Administration of Injectable PEG-Irinotecan (JK-1201I) in Patients with Malignant Solid Tumor
Brief Title: Safety, Tolerability and Pharmacokinetics of Injectable PEG-Irinotecan (JK-1201I) in Patients with Malignant Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JenKem Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: JK-1201I-P1
Record Dates: First submitted 2020-04-08; First posted 2020-04-29 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open labled, positive controled, single, -combined, with multiple dose escalation trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- 50mg/m2 (Experimental): Starting dose, administered once only
  Interventions: Drug: JK-1201I
- 75mg/m2 (Experimental): Second dose level, administered at least twice, first two cycles of drug delivery accompanied with PK analyses.
  Interventions: Drug: JK-1201I
- 100mg/m2 (Experimental): Third dose level, administered at least twice, first two cycles of drug delivery accompanied with PK analyses.
  Interventions: Drug: JK-1201I
- 125mg/m2 (Experimental): Forth dose level, administered at least twice, first two cycles of drug delivery accompanied with PK analyses.
  Interventions: Drug: JK-1201I
- 150mg/m2 (Experimental): Fifth dose level, administered at least twice, first two cycles of drug delivery accompanied with PK analyses.
  Interventions: Drug: JK-1201I
- 180mg/m2 (Experimental): Sixth dose level, administered at least twice, first two cycles of drug delivery accompanied with PK analyses.
  Interventions: Drug: JK-1201I
- 175mg/m2 (Active Comparator): CPT-11, given every 14 days, first 2 cycles of drug delivery will accompanied with PK test,
  Interventions: Drug: JK-1201I

INTERVENTIONS:
Drug: JK-1201I — malignant solid tumor that has been confirmed by histopathology and/or cytology

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of injectable PEG-Irinotecan in patients with malignant solid tumors

DETAILED DESCRIPTION:
This study is a multicenter, open labeled, positive controlled, single, -combined, with multiple dose escalation trial.

The trial consists of 6 drug dose groups, which are 50mg/m2, 75mg/m2, 100mg/m2, 125mg/m2, 150mg/m2 and 180mg/m2 respectively. At each testing dose group, one patient will be treated with HCl-Irinotecan (CPT-11), at dose level of 175mg/m2.

The initial dose of 50mg /m2 will be administered once. Starting from the 75mg/m2 dose group, each patient will be given testing drug at least twice. During first and second drug administration, blood samples will be collected for PK characteristics analysis. Patients will be evaluated after every two rounds of drug delivery and preliminary efficacy of testing compound will be determined as PD, SD, CR etc.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years of age (inclusive)；
2. Body mass index (BMI) within the range of 19-30 (inclusive)
3. Patient with a malignant solid tumor that has been confirmed by histopathology and/or cytology to be ineffective in conventional treatment or lack effective treatment。 Primary tumors include colorectal cancer, gastric cancer, esophageal cancer, pancreatic cancer and advanced breast cancer patients with brain metastases
4. More than 4 weeks after the completion of previous anti-tumor therapy (including chemotherapy/radiotherapy, surgical treatment, targeted therapy, immunotherapy, Chinese herbal medicine therapy, endocrine therapy or other anti-tumor therapy), And it has recovered from the adverse reactions of previous treatments (treatment-related toxicity grade ≤1);
5. At least one measurable or evaluable lesion was identified using RECIST 1.1;
6. Physical state score (ECOG PS score) 0~1
7. Estimated survival time ≥ 3 months
8. Both standard blood tests and Blood Biochemistry tests are within normal range.
9. All subjects and their partners have no plan to have children from screening to 6 month after the trial, and those who agree to use effective non-drug contraceptive methods during the trial period (e.g., condoms， etc.), those already have permanent contraceptive measures, such as bilateral tubal ligation, vasectomy, etc.
10. Voluntarily participate in clinical research and sign informed consent

Exclusion Criteria:

1. Patients with previous allergy history and known severe allergy to injectable PEG-Irinotecan or any excipient of the product;
2. Have received HCl-Irinotecan (CPY-11) treatment in the past
3. With active brain metastasis;
4. Have other malignant tumors within 5 years before enrollment, except for previously treated with the purpose of radical cure such as carcinoma in situ of the cervix, squamous cell carcinoma or basal cell carcinoma
5. Large amount of thorax and ascites that need treatment
6. Serious cardiovascular disease, including grade II and above cardiac dysfunction (NYHA standard)
7. Active hepatitis b (HBsAg and/or HBCAb positive, peripheral blood HBV DNA titer test ≥1×103 IU/mL, or hepatitis c patients; or testing positive for syphilis or human immunodeficiency virus (HIV);
8. Subject is participating in other clinical studies or the presumed first time of drug administration is less than 4 weeks from the end of the previous clinical study (last administration or 5 half-lives of the previous study drug);
9. Subjects who have been treated with anti-tumor vaccines or other anti-tumor drugs (interferon, interleukin, etc.) with immune-stimulatory effects within 28 days before the assumed first medication
10. Subjects who had a severe infection within 4 weeks before the first medication， including but not limited to complications of infection, bacteremia, severe pneumonia and others requiring hospital stays;
11. Patient has electrolyte disorder with clinically significance
12. Subject has clinically severe gastrointestinal disorders, (positive fecal occult blood with severe gastrointestinal bleeding, gastrointestinal infection, obstruction or diarrhea of grade 1 or above on endoscopic examination (the number of stool increases ≥4 times per day))
13. Patients with bleeding tendency or receiving thrombolytic or anticoagulant therapy
14. Within 14 days before receiving the study drug treatment subject have used a strong CYP3A4 inducer (Phenytoin or Carbamazepine, Barbiturates, Rifampicin or Rifabutin, Hypericum perforatum, etc.);
15. Within 7 days prior drug treatment, patients have used strong CYP3A4 inhibitors (Clarithromycin, Ketoconazole or Itraconazole, Indinavir, Lopinavir, Nafazodone, Nelfinavir, Ritonavir, Saquinavir, Trapavir, Voriconazole, etc.)
16. Within 7 days before receiving study drug treatment, subject has used strong UGT1A1 inhibitors (Atazanavir, Gemfibrozil, etc.)
17. Clear history of neuropathy or mental disorders (including epilepsy or dementia)
18. Persons with a history of alcohol or drug abuse
19. Pregnant or lactating women
20. Investigator considered the subject who are not suitable to participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome 1 | 21 days
  Maximum tolerance dose (MTD) will be determined. MTD is defined as the highest dose that can be given without causing any adverse side effects according to CTCAE v5.0.
  The dose climbing scheme was designed according to the improved Fibonacci method, which was carried out in sequence from the low dose group to the high dose group. The principle of "3+3" dose increment was adopted. At least 4 subjects were randomly enrolled in each dose group (including one patient who will be assigned to control drug).
Primary outcome 2 | 21 days
  Dose limited toxicity (DLT) of injectable PEG -Irinotecan in patients will be determined.
  DLT is defined as: 1..Grade 4 neutropenia (ANC) reduction lasts ≥3 days; or grade 3 ANC reduction with fever (ANC <1000 / mm3 with oral temperature single measurement> 38.3 ℃ or ≥38.0 ℃ for 1 hour)； 2. Grade 3 thrombocytopenia (25×109/L≤ platelet count < 50×109/L) with obvious clinical bleeding symptoms, or grade 4 thrombocytopenia (with or without obvious clinical bleeding symptoms); 3. Other grade 4 hematological toxicity； 4. Grade 3 and above non-hematological toxicity； 5. Hair loss, fatigue, except for those with grade 3 nausea, vomiting, and diarrhea without maximum symptomatic supportive treatment.

SECONDARY OUTCOMES:
Secondary outcome 1 | 21 days
  Serum concentration of injectable PEG-Irinotecan , Irinotecan and SN-38 in human subjects.
  Blood samples will be taken within 60min before administration, 10min±5min after intravenous infusion, 10min±5min before the end of intravenous infusion, immediately after intravenous infusion 0h±5min, thereafter 15min±5min, 30min±5min, 1h±5min, 2h±10min, 4h±15min, 8h±30min, 12h±30min, 24h±1h, 48h±2h, 72h±2h, 96h±2h, 168h±2h; A total of 16 time points were collected in each patient. The concentrations of PEG-Irinotecan, irinotecan and the active metabolite SN-38 will be determined by LC-MS/MS. And the maximum concentration (Cmax) and the time of peak of concentration (Tmax) will be compared across different groups.
Secondary outcome 2 | 21 days
  Objective Response Rate (ORR) of injectable PEG-Irinotecan in patients. Per Response Evaluation Criteria In Solid Tumors (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhao, Ph.D., Study Chair — JenKem Technology Co., Ltd.
Locations (1):
- The fifth medical center of PLA general hospital, Beijing, Beijing Municipality, China